CLINICAL TRIAL: NCT03374878
Title: E5 - Oral Contraceptive and Strength Training (2nd Generation)
Brief Title: Oral Contraceptive and Strength Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Mette Hansen, Associate Professor, University of Aarhus
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: VEK60597
Record Dates: First submitted 2017-12-05; First posted 2017-12-15 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2018-06

CONDITIONS: Healthy
Keywords: exercise; oral contraceptive; strength training
MeSH Terms: conditions — Motor Activity | interventions — Contraceptives, Oral

STUDY DESIGN:
Intervention Model Description: Cross sectional study with 16 in each group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oral contraceptive and training (Experimental): Users of oral contraceptive training for 10 weeks
  Interventions: Other: oral contraceptive and training
- no oral contraceptive and training (Placebo Comparator): Non-users of oral contraceptive training for 10 weeks
  Interventions: Other: no oral contraceptive and training

INTERVENTIONS:
Other: no oral contraceptive and training — 10 weeks of training in a group of oral contraceptive users
  Arms: no oral contraceptive and training
Other: oral contraceptive and training — 10 weeks of training in a group of users of oral contraceptives
  Arms: oral contraceptive and training

SUMMARY:
Cross sectional study investigating the effect of strength training in users and non-users of oral contraceptives (OC) (2nd generation OC)

ELIGIBILITY:
Inclusion Criteria:

* 18.5 - 30 years
* BMI < 30

Exclusion Criteria:

* Medicine influencing protein turnover
* Surgery on the knee
* Arthritis
* Diabetes
* Smoking
* irregular menstruation (<24 days or >35 days cycles)
* Non-users: not have used contraceptives for the last 3 months.
* Unstable weight (+/- 5 kg within the last 6 months)
* Regular training/exercise more than 2 hours/week for the last 6 months. Maximum 70 km of cycling transport/week.
* Strength training >1time/month for the last 6 months.
* Pregnancy
* Diet og eating disorder
* Can not read or understand danish

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Use of oral contraceptives compared to same sex controls.
Enrollment: 38 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Muscle mass | Baseline + after 10 weeks of resistance training.
  Change in muscle mass determined by MRI scan of thigh muscle

SECONDARY OUTCOMES:
Muscle fiber size | Baseline + after 10 weeks of resistance training.
  Change in muscle fiber cross sectional area measured by histology.
Muscle strength | Baseline + after 10 weeks of resistance training.
  Change in isometric strength
Blood values | Baseline + after 10 weeks of resistance training.
  Change in sex hormone profile measured by blood sample analysis
Functionality | Baseline + after 10 weeks of resistance training.
  Change in jump performance by RSI (Reactive strength index) measures
Fat free mass (FFM) | Baseline + after 10 weeks of resistance training.
  Change in FFM measured by dual energy x-ray absorptiometry (DXA) scan of whole body composition

CONTACTS AND LOCATIONS:
Overall Officials: Mette Hansen, PhD, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University, Department for Public Health, Section for Sport Science, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No